CLINICAL TRIAL: NCT04595500
Title: Gastroesophagial Reflux Disease as a Potential Contributor to Dental Erosions and Oral Tissue Alterations
Brief Title: Relationship Between Gastroesophageal Reflux Disease and Dental Erosion
Status: Completed | Type: Observational
Sponsor: University of Beykent (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Fatma AYTAC BAL, Assistant professor, University of Beykent
Other Study IDs: 131/2-2008
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Gastroesophageal Reflux Disease; Tooth Wear
Keywords: Dental erosion; DMFT; Gastroesophageal Reflux Disease; Saliva
MeSH Terms: conditions — Gastroesophageal Reflux; Tooth Wear; Tooth Erosion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GERD
- Control

SUMMARY:
This study aimed to investigate the relationship between gastroesophageal reflux disease (GERD) and dental erosion and the alterations in oral tissues. This was a case-control study. The GERD group consisted of 50 individuals with endoscopic esophagitis who had gastroesophageal reflux symptoms, and the control group consisted of 50 healthy individuals. The prevalence of teeth wear and caries was evaluated using the Smith and Knight tooth wear index (TWI) and the decayed, missing, and filled teeth index (DMFT), respectively. Inflammatory mouth sensitivity, tongue sensitivity, nonspecific itching and burning, halitosis, dry mouth, teeth sensitivity, and the erythema of the soft and hard palatal mucosa and uvula were also evaluated. Stimulated saliva samples were collected, and the salivary flow rate, pH, and buffering capacity values were measured.

ELIGIBILITY:
Inclusion Criteria:

* The patient group included with at least one year of reflux symptoms, endoscopic esophagitis, no systemic disease other than reflux, no medication use except anti-reflux drugs, no habit of ruminating and vomiting, and no habit of bruxism.
* The control group included without any systemic disorder, no habit of ruminant and vomiting, no habit of bruxism, and no drug use.

Exclusion Criteria:

* The volunteers who were vegetarian, consumed citrus and vinegar frequently, and consumed more than ½ liter of acidic beverages per day were not included in the study. Those who never brush their teeth and were using battery/rechargeable and scrub brush and abrasive toothpaste were not included in the study, either.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This case-control study was conducted in Ankara University Faculty of Dentistry, Department of Restorative Dentistry Polyclinics and Ankara University Faculty of Medicine, Department of Gastroenterology Polyclinics with a total of 100 participants (49 females and 51 males between the ages of 16-65) of whom 50 were in the GERD group, and 50 were in the control group. Among the patients who were admitted to the clinics, those with a diagnosis of GERD were included in the patient group and those without GERD were included in the control group. Ethical approval of the study protocol was granted by the Ankara University Faculty of Dentistry Research Ethics Committee (No:131/2 Date:10.06.2008).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
TWI (Smith and Knight tooth wear index) | Baseline
  Score 0 No loss of enamel surface characteristics. No loss of contour. Score 1 Loss of enamel surface characteristics. Minimal loss of contour. Score 2 Loss of enamel exposing dentine for less than one third of surface. Loss of enamel just exposing dentine. Defect less than 1 mm deep.
  Score 3 Loss of enamel exposing dentine for more than one third of surface. Loss of enamel and substantial loss of dentine. Defect less than 1-2 mm deep.
  Score 4 Complete enamel loss - pulp exposure - secondary dentin exposure. Pulp exposure or exposure of secondary dentine. Defect more than 2mm deep - pulp exposure - secondary dentine exposure.
DMFT index | Baseline
  The decayed, missing, and filled teeth index
Salivary flow rate | Baseline
  Saliva collection was performed between 9:00 and 12:00 in the morning. Stimulation for the collection of saliva samples was provided by sugar-free gum. Saliva flow rate was recorded as ml / min by dividing the amount obtained after 5 minutes of chewing by the time.
pH value | Baseline
  The pH value of saliva samples was measured with a pH meter (Sentron digital pH-meter, Nisan Inc.,Turkey). The calibration procedure of the device was done in accordance with the manufacturer's instructions and using standard pH buffers.
Buffering capacity | Baseline
  The buffering capacity of the collected saliva samples was determined according to the Ericsson method.The collected stimulated saliva was taken into another sterile glass tube by drawing 1 ml without waiting. 3ml 0.005 N HCl was added onto it and the vessel was vibrated slightly to remove carbon dioxide and the pH value was measured with a pH meter (Sentron digital pH-meter, Nisan Inc.,Turkey).
Oral complaints | Baseline
  Oral complaints of the participants were evaluated according to the answers given to the questions regarding inflammatory mouth sensitivity, tongue sensitivity, nonspecific itching and burning in the mucosa, halitosis, dry mouth, and increased teeth sensitivity. The presence of erythema in the soft/hard palatal mucosa/uvula was determined by oral examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Aytac Bal, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes